CLINICAL TRIAL: NCT02608801
Title: Prediction and Secondary Preventing of Fractures in a Norwegian Population. A Substudy of Norwegian Capture the Fracture Initiative
Brief Title: Prediction and Secondary Prevention of Fractures
Acronym: NOFRACTsub
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Asker & Baerum Hospital (Other); Drammen sykehus (Other); Haukeland University Hospital (Other); Molde Hospital (Other); Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Frede Frihagen, Consultant, Oslo University Hospital
Other Study IDs: 2014/2260REK OS
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Osteoporotic Fractures; Hip Fractures; Wrist Fractures; Ankle Fractures; Vertebral Compression Fractures; Humeral Fractures, Proximal
MeSH Terms: conditions — Osteoporotic Fractures; Hip Fractures; Wrist Fractures; Ankle Fractures; Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients from NoFRACT: Patients from NoFRACT who consent to participate in this sub-study, will be offered examination and treatment with anti-osteoporotic drugs cf. treatment algorithm in the main-study. I.e. if osteoporosis is present clinically or at DXA scan, treatment is started.

SUMMARY:
The purpose of this study is to investigate patient related factors that contribute to increased risk of recurrent fractures and to investigate patient adherence to prescribed anti-osteoporotic drugs.

DETAILED DESCRIPTION:
A standardized treatment program of osteoporosis will be introduced successively at 7 hospitals in Norway from April 2015 to January 2016. This Project is named NoFRACT (Norwegian Capture the Fracture Initiative https://clinicaltrials.gov/show/NCT02536898). Patients above 50 years of age, who recently have suffered a fragility fracture, will be offered examination of osteoporosis and treatment if indicated. Some of these patients will be asked to participate in this consent-based sub-study (NoFRACTsub). At baseline, the patients will be asked to answer a questionnaire, collect blood-sample for to outline possible causes for osteoporosis, in addition to Dual X-Ray Apsopiometry (DXA) scan including bone mineral density(BMD), trabecular bone score(TBS) and vertebral fracture assessment (VFA). At 1-year follow-up there will be a brief questionnaire and measuring of BTM. At 2-year follow-up there will be a brief questionnaire in addition to repeated measurement of DXA including BMD, TBS and VFA. All data will be stored securly at the designated server at the University of Oslo, Service of sensitive data, TSD.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in NoFRACT
* Recent low-trauma vertebral or non-vertebral fracture
* Written patient consent

Exclusion Criteria:

* Fractures of scull, face, toes or fingers
* Short life expectancy
* Patients not competent or willing to give consent
* Patients having difficulties in answering questionairies, undergoing a DXA scan, and show up on the follow-ups,

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already enrolled in NoFRACT main-study. Some patients will be asked to participate in this consent based sub-study, and must be able to answer questionairies, undergo DXA scan and bloodtests at baseline and follow-up.
Sampling Method: Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Fragility fractures | 2 years
  Number of new fractures during observation periode

SECONDARY OUTCOMES:
Bone mineral Density (BMD) | Baseline, 2 years
  BMD in g/cm2 measured by DXA at both hips and lumbar spine. We want to study if there is a correlation between BMD an incidence of new fractures
Trabecular Bone Score (TBS) | Baseline, 2 years
  TBS is an absolute value calculated from the DXA scans of L1-L4. We want to see if TBS can be used as a predictor of future fractures
Spinal Deformity Index (SDI) | Baseline, 2 years
  Grading of vertebral fractures (SQ1=1 point, SQ2 =2 points, SQ3= 3 points) by Vertebral Fracture Assessment of lateral DXA scans. The total of points is the SDI. We want to see if there is a correlation between present fractures at baseline and future fractures
s-CTX | At 1 year follow-up
  Fasting CTX (carboxy-terminal collagen crosslinks)in serum, measured in pg/ml
s-PINP | At 1 year follow-up
  Fasting PINP (Procollagen I Intact N-Terminal)in Serum, measured in mcg/L
FRAX score | Baseline
  Calculation 10-year fracture risk for major osteoporotic and hip fractures by FRAX calculated during DXA scanning, on a population treated with AOD
Garvan score | Baseline
  Calculation of 10-year fracture risk for major osteoporotic and hip fracture using online available Garvan Nomogram, on a population treated with AOD.
Self-reported adherence to anti-osteoporotic drugs (AOD) | Baseline, 1 year, 2 years
  Self-reported use of AOD by questionnaire. Answer yes or no. If terminating of the treatment, patients will be asked to describe why.

CONTACTS AND LOCATIONS:
Overall Officials: Åshild Bjørnerem, Dr Med, Study Director — The Arctic University of Norway
Locations (6):
- Norway (6):
  - Baerum Hospital, Sandvika, Gjettum
  - St. Olavs Hospital, Trondheim, Trønderlag
  - Drammen hospital, Drammen
  - Molde Hospital, Molde
  - Orthopedic Center, Ulleval University Hospital, Oslo
  - University Hospital of North Norway, Tromsø

REFERENCES:
- See also: NoFRACT — https://clinicaltrials.gov/show/NCT02536898